CLINICAL TRIAL: NCT02253316
Title: A Phase II Study of IRD (Ixazomib, Lenalidomide, & Dexamethasone) for Consolidation Therapy Post Autologous Stem Cell Transplantation Followed by Maintenance Ixazomib or Lenalidomide for Multiple Myeloma
Brief Title: Phase II Study of IRD (Ixazomib, Lenalidomide, Dexamethasone) Post Autologous Stem Cell Transplantation Followed by Maintenance Ixazomib or Lenalidomide for Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Multiple Myeloma Research Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201411060
Record Dates: First submitted 2014-09-24; First posted 2014-10-01 (Estimated); Results first posted 2021-09-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Autologous Stem Cell Transplantation; Ixazomib; Lenalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone; Calcium Dobesilate; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Consolidation: Ixazomib, Lenalidomide, & Dexamethasone (Experimental): Consolidation therapy will begin between Day 80 and Day 120 following ASCT and will consist of four 28-day cycles of IRD (ixazomib, lenalidomide, & dexamethasone). Barring dose modifications for toxicity, 4 mg of ixazomib and 40 mg of dexamethasone will be administered on Days 1, 8, and 15, and 15 mg of lenalidomide will be administered on daily on Days 1-21.
  Interventions: Biological: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone
- Maintenance Arm 1: Ixazomib (Experimental): Ixazomib will be administered on Days 1, 8, and 15 of a 28-day cycle at a starting dose of 4 mg until patient progresses or experiences an unacceptable toxicity.
  Interventions: Biological: Ixazomib
- Maintenance Arm 2: Lenalidomide (Experimental): Lenalidomide will be administered daily continuously for a 28-day cycle at a starting dose of 10 mg. If lenalidomide is tolerated well (i.e. no dose modification required) during the first three cycles, lenalidomide dose will be increased to 15 mg daily and will continue until patient progresses or experiences an unacceptable toxicity.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Biological: Ixazomib
  Other Names: [14C]-ixazomib; [14C]-MLN9708
  Arms: Consolidation: Ixazomib, Lenalidomide, & Dexamethasone; Maintenance Arm 1: Ixazomib
Drug: Lenalidomide
  Other Names: Revlimid
  Arms: Consolidation: Ixazomib, Lenalidomide, & Dexamethasone; Maintenance Arm 2: Lenalidomide
Drug: Dexamethasone
  Other Names: Aeroseb-Dex; Alba-Dex; Decaderm; Decadrol; Decadron; Decasone R.p.; Decaspray; Deenar; Deronil; Dex-4; Dexace; Dexameth; Dezone; Gammacorten; Hexadrol; Maxidex; Sk-Dexamethasone
  Arms: Consolidation: Ixazomib, Lenalidomide, & Dexamethasone

SUMMARY:
The purpose of this research study is to evaluate a treatment regimen called IRD which will be given to participants after their stem cell transplant in an effort to help prolong the amount of time the participants are disease-free after transplant. IRD is a three-drug regimen consisting of ixazomib, lenalidomide (also called Revlimid), and dexamethasone. After 4 cycles of IRD, the participants will be randomized to receive maintenance therapy either with ixazomib or lenalidomide.

DETAILED DESCRIPTION:
Based on the further need to improve progression-free survival and overall survival post-autologous stem cell transplantation (ASCT) for multiple myeloma and the benefits seen of consolidation/maintenance treatment with immunomodulatory drugs thalidomide and lenalidomide and the proteasome inhibitor bortezomib, the natural next step is to evaluate combination regimens of immunomodulatory drugs and proteasome inhibitors as consolidation/maintenance post-ASCT. The regimen consisting of ixazomib, lenalidomide, and dexamethasone (IRD) has been shown to have low toxicity, and the availability of an oral formulation of ixazomib allows for easier administration when compared to bortezomib.

In this study, following consolidation with IRD, patients will be randomized to maintenance therapy with lenalidomide or ixazomib in order to collect pilot data comparing the toxicity and efficacy of maintenance therapy with immunomodulatory drugs and proteasome inhibitors.

09/23/2019: Upon review of the interim analysis, there will be no further randomizations into the maintenance portion of the trial. All patients will be enrolled into the lenalidomide arm with the exception of those who discontinue lenalidomide during the consolidation phase due to toxicity. Patients who discontinue lenalidomide may be enrolled into the ixazomib arm following approval from the principal investigator.

09/30/2021: Following analysis 4 in 2021, analysis of the primary endpoint, all patients receiving lenalidomide maintenance will be transitioned off-study. Patients receiving ixazomib may remain on trial until disease progression or unacceptable toxicity at the discretion of the treating physician and the site principal investigator.

ELIGIBILITY:
Inclusion Criteria

Each patient must meet all of the following inclusion criteria to begin IRD Consolidation:

* Between the ages of 18 and 70 years of age (inclusive) at time of enrollment
* Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Confirmed diagnosis of symptomatic multiple myeloma. (Patients with multiple myeloma with secondary amyloidosis are eligible.)
* Received at least two cycles of any regimen as initial systemic therapy for multiple myeloma and are within 2-16 months of the first dose of initial therapy
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2
* Adequate organ function as defined below:

Absolute neutrophil count (ANC) >= 1,000 mm^3 Platelet count >= 75,000/mm^3; platelet transfusions to help patient meet eligibility criteria are not allowed within 7 days before study enrollment Total bilirubin <= 1.5 x upper limit of normal range (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=3 x ULN Calculated creatinine clearance >= 30 mL/min

* Women of childbearing potential must follow pregnancy testing requirements as outlined in the Revlimid REMS program material. This is defined as either committing to continued abstinence from heterosexual intercourse or beginning TWO acceptable methods of contraception (one highly effective method and one additional effective method AT THE SAME TIME) at least 28 days prior to the start of lenalidomide, for the duration of study participation, and for 28 days following the last dose of lenalidomide. Women of childbearing potential must also agree to ongoing pregnancy testing.
* Men must agree to use a latex condom during sexual contact with a woman of childbearing potential even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* All study participants must be registered into the mandatory Revlimind REMS program and be willing to comply with its requirements. Per standard Revlimid REMS program requirements, all physicians who prescribe lenalidomide for research subjects enrolled into this trial, must be registered in, and must comply with, all requirements of the Revlimid REMS program.

Exclusion Criteria

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Evidence of MM disease progression any time prior to enrollment. Progression from smoldering/asymptomatic MM to symptomatic MM is not exclusionary.
* Tandem autologous transplantation
* History of plasma cell leukemia or MM CNS involvement
* Administration or planned administration of any other concomitant chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy which would be considered a treatment of multiple myeloma until Day +28 post-transplant through discontinuation from study. Patients may be on corticosteroids if they are being given for disorders other than multiple myeloma (e.g., adrenal insufficiency, rheumatoid arthritis, etc.)
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Prior organ transplant requiring immunosuppressive therapy
* Active hepatitis A, B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib
* Concurrent hematologic or non-hematologic malignancy requiring treatment (other than multiple myeloma and secondary amyloidosis)
* Cardiac syncope, uncompensated NYHA Class 3 or 4 congestive heart failure, myocardial infarction within the previous six months, unstable angina pectoris, clinically significant repetitive ventricular arrhythmias despite antiarrhythmic treatment, severe orthostatic hypotension, or clinically important autonomic disease
* Grade >= 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period
* Major surgery within 14 days prior to enrollment
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days prior to enrollment
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days prior to enrollment and throughout the duration of this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2026-08-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (10):
- United States (10):
  - City of Hope, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Tennessee Oncology, PLLC, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Maintenance Arm 1: Ixazomib: Ixazomib will be administered on Days 1, 8, and 15 of a 28-day cycle at a starting dose of 4 mg until patient progresses or experiences an unacceptable toxicity.
  09/23/2019: Upon review of the interim analysis, there will be no further randomizations into the maintenance portion of the trial. All patients will be enrolled into the lenalidomide arm with the exception of those who discontinue lenalidomide during the consolidation phase due to toxicity. Patients who discontinue lenalidomide may be enrolled into the ixazomib arm following approval from the principal investigator.
Period: Consolidation
Arm/Group | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone | Maintenance Arm 1: Ixazomib | Maintenance Arm 2: Lenalidomide
Started | 236 | 0 | 0
Completed | 220 | 0 | 0
Not Completed | 16 | 0 | 0
Not completed — Progression | 4 | 0 | 0
Not completed — Non-Compliance | 1 | 0 | 0
Not completed — Patient Withdrew Logistical Concerns | 2 | 0 | 0
Not completed — Secondary Malignancy | 2 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0
Period: Maintenance
Arm/Group | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone | Maintenance Arm 1: Ixazomib | Maintenance Arm 2: Lenalidomide
Started | 0 | 99 | 116
Completed | 0 | 70 | 74
Not Completed | 0 | 29 | 42
Not completed — Patient Withdrew Logistical Concerns | 0 | 7 | 7
Not completed — Physician Decision | 0 | 7 | 16
Not completed — Non-Compliance | 0 | 1 | 1
Not completed — Secondary Malignancy | 0 | 2 | 6
Not completed — Adverse Event | 0 | 8 | 12
Not completed — Still receiving active treatment | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone
Number analyzed (Participants) | 236
Age, Continuous [Median (Full Range); unit: years] | 58 [28 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 217
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 185
  More than one race | 1
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 236

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement in Minimal Residual Disease (MRD)
Description: For the purposes of this study, a patient will be considered as having minimal residual disease if a positive result (1x10E06) is obtained using the Adaptive Clonoseq MRD testing.
Time Frame: After 4 cycles of IRD consolidation treatment (approximately Day 112 of consolidation treatment)
Population: Only participants in the consolidation portion of the trial are evaluable for this outcome measure. 52 patients in consolidation were not evaluable for the outcome because 26 did not have appropriate VDJ rearrangements on clonoSEQ assessment, 10 did not have sample available from one or both time points, and 16 were removed prior to completion of 4 cycles of IRD.
Measure: Count of Participants; unit: Participants
Arm/Group | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone | Maintenance Arm 1: Ixazomib | Maintenance Arm 2: Lenalidomide
Number analyzed (Participants) | 184 | 0 | 0
Participants | 19 |  |

2. Secondary Outcome: MRD-negative Rate After ASCT
Description: as for outcome 1
Time Frame: Prior to beginning consolidation treatment (Day -28 to Day 0)
Population: Only participants in the consolidation portion of the trial are evaluable for this outcome measure. 33 patients from consolidation were not evaluable for this outcome because 26 patients did not have appropriate VDJ rearrangements found on clonSEQ assessment and 7 patients did not have a sample available.
Measure: Count of Participants; unit: Participants
Arm/Group | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone | Maintenance Arm 1: Ixazomib | Maintenance Arm 2: Lenalidomide
Number analyzed (Participants) | 203 | 0 | 0
Participants | 51 |  |

3. Secondary Outcome: Toxicity of IRD Consolidation
Description: For the purposes of this study, toxicity will be defined as inability to receive 4 cycles of IRD consolidation due to toxicity.
Time Frame: After 4 cycles of IRD consolidation treatment (approximately Day 112 of consolidation treatment)
Population: Only participants in the consolidation portion of the trial are evaluable for this outcome measure. 10 patients in consolidation were not evaluable for this outcome because they discontinued prior to 4 cycles of IRD for reasons other than toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone | Maintenance Arm 1: Ixazomib | Maintenance Arm 2: Lenalidomide
Number analyzed (Participants) | 226 | 0 | 0
Participants | 7 |  |

4. Secondary Outcome: Response Rate of IRD Consolidation
Description: For the purposes of this study, response rate is defined as the improvement in complete response rate. Response will be determined by the International Myeloma Working Group (IMWG) Uniform Response Criteria.
Time Frame: After 4 cycles of IRD consolidation treatment (approximately Day 112 of consolidation treatment)
Population: Only participants in the consolidation portion of the trial are evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone | Maintenance Arm 1: Ixazomib | Maintenance Arm 2: Lenalidomide
Number analyzed (Participants) | 236 | 0 | 0
Participants | 49 |  |

5. Secondary Outcome: Progression-free Survival of IRD Consolidation
Description: Progression-free survival (PFS) will be defined as time from ASCT to progression, relapse, or death, whichever occurs first, and those event-free survivors will be censored at withdrawal or study closeout.
Time Frame: Up to 18 months after completion of maintenance therapy (Up to 5 years after starting the study)
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival of IRD Consolidation
Description: Overall survival (OS) will be defined as time from ASCT to death due to any causes, and survivors will be censored at withdrawal or study closeout.
Time Frame: Up to 18 months after completion of maintenance therapy (Up to 5 years after starting the study)
Reporting Status: Not Posted

7. Secondary Outcome: Compare Toxicity Between the Two Maintenance Arms
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Time Frame: 30 days after the completion of maintenance treatment (estimated to be Day 1125 of maintenance treatment)
Reporting Status: Not Posted

8. Secondary Outcome: Compare Response Rate Between the Two Maintenance Arms
Description: * Response will be determined by the International Myeloma Working Group (IMWG) Uniform Response Criteria. Response includes stringent complete response (sCR) and complete response (CR).
  * sCR requires all of the following:
    * CR as defined below
    * Normal free light chain ratio (0.26-1.65)
    * Absence of clonal cells in the bone marrow by immunohistochemistry or immunofluorescence
  * CR requires all of the following:
    * Disappearance of monoclonal protein by both protein electrophoresis and immunofixation studies from the blood and urine
    * If serum and urine monoclonal protein are unmeasurable, Normal free light chain ratio (0.26-1.65)
    * <5% plasma cells in the bone marrow
    * Disappearance of soft tissue plasmacytoma
Time Frame: Through completion of maintenance treatment (estimated to be day 1095 of maintenance treatment)
Population: This outcome measure is only for participants who went onto the maintenance arms. Participants in the maintenance arms were not evaluable for this outcome measure if they were removed from treatment for reasons other than progressive disease prior to Month 13.
Measure: Count of Participants; unit: Participants
Arm/Group | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone | Maintenance Arm 1: Ixazomib | Maintenance Arm 2: Lenalidomide
Number analyzed (Participants) | 0 | 91 | 109
Participants |  | 50 | 80

9. Secondary Outcome: Compare Progression-free Survival Between the Two Maintenance Arms
Description: as for outcome 5
Time Frame: Up to 18 months after completion of maintenance therapy (Up to 5 years after starting the study)
Reporting Status: Not Posted

10. Secondary Outcome: Compare Overall Survival Between the Two Maintenance Arms
Description: as for outcome 6
Time Frame: Up to 18 months after completion of maintenance therapy (Up to 5 years after starting the study)
Reporting Status: Not Posted

11. Secondary Outcome: Rate of MRD-positive to MRD-negative Conversion Between the Two Maintenance Arms
Time Frame: Cycle 13 Day 1 of maintenance treatment (Approximately Day 364 of maintenance treatment)
Population: This outcome measure is only for participants who went onto the maintenance arms. For the maintenance arms, the overall number of participants analyzed only includes those participants who were MRD positive at the start of maintenance.
Measure: Count of Participants; unit: Participants
Arm/Group | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone | Maintenance Arm 1: Ixazomib | Maintenance Arm 2: Lenalidomide
Number analyzed (Participants) | 0 | 57 | 52
Participants |  | 5 | 11

12. Secondary Outcome: Association of Progression-free Survival With MRD-negativity
Description: as for outcome 5
Time Frame: Up to 18 months after completion of maintenance therapy (Up to 5 years after starting the study)
Reporting Status: Not Posted

13. Secondary Outcome: Association of Progression-free Survival With MRD-positivity
Description: as for outcome 5
Time Frame: Up to 18 months after completion of maintenance therapy (Up to 5 years after starting the study)
Reporting Status: Not Posted

14. Secondary Outcome: Association of Overall Survival With MRD-negativity
Description: as for outcome 6
Time Frame: Up to 18 months after completion of maintenance therapy (Up to 5 years after starting the study)
Reporting Status: Not Posted

15. Secondary Outcome: Association of Overall Survival With MRD-positivity
Description: as for outcome 6
Time Frame: Up to 18 months after completion of maintenance therapy (Up to 5 years after starting the study)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: -Adverse events were collected from first dose of study treatment through 30 days after the completion of study treatment. -All-cause mortality time frame is from first dose of study treatment through 30 days after the completion of study treatment.
Arm/Group | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone | Maintenance Arm 1: Ixazomib | Maintenance Arm 2: Lenalidomide
All-Cause Mortality (participants affected / at risk) | 1/236 | 0/99 | 1/116
Serious Adverse Events (participants affected / at risk) | 44/236 | 24/99 | 48/116
Other Adverse Events (participants affected / at risk) | 236/236 | 99/99 | 116/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone (N=236) | Maintenance Arm 1: Ixazomib (N=99) | Maintenance Arm 2: Lenalidomide (N=116)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Coronary artery calcification (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 2 | 2
Chloecystitis (Hepatobiliary disorders) | 0 | 0 | 4
Anaphylaxis - shellfish (Immune system disorders) | 0 | 0 | 1
C. difficile infection (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 12 | 2 | 12
Salmonella enteritis infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 1
Skin infection (Infections and infestations) | 0 | 1 | 1
Upper respiratory infection (Infections and infestations) | 8 | 12 | 10
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Ixazomib overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pancytopenia (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute lymphoblastic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer in Situ (DCIS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Compression fracture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papillary urothelial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Plasmacytoma (myeloma progression) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Spinal cord compression (myeloma progression) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 5
Tubulovillous adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1
Neuropathic back pain (Nervous system disorders) | 1 | 0 | 0
Ocular migraine (Nervous system disorders) | 0 | 1 | 0
Rigors (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Altered mental status (Psychiatric disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Renal calculi (Renal and urinary disorders) | 0 | 0 | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Consolidation: Ixazomib, Lenalidomide, & Dexamethasone (N=236) | Maintenance Arm 1: Ixazomib (N=99) | Maintenance Arm 2: Lenalidomide (N=116)
Anemia (Blood and lymphatic system disorders) | 120 | 44 | 60
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Hemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 1 | 1
Arrhythmia NOS (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 3 | 0 | 2
Heart murmur (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 3 | 1 | 3
Sinus bradycardia (Cardiac disorders) | 2 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 3 | 1 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 4
Eustachian tube disfunction (Ear and labyrinth disorders) | 1 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 2 | 2
Middle ear inflammation (Ear and labyrinth disorders) | 3 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 2 | 4
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 3
Cushingoid (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Hypoparathyroidism (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 2 | 1
Thyroiditis (Endocrine disorders) | 0 | 0 | 1
Allergic eye irritation (Eye disorders) | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1
Blurred vision (Eye disorders) | 10 | 9 | 8
Bulging retinas (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0
Conjuctivitis (Eye disorders) | 3 | 0 | 2
Dry eye (Eye disorders) | 3 | 4 | 1
Eye pain (Eye disorders) | 2 | 1 | 1
Floaters (Eye disorders) | 0 | 2 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Itchy eyes (Eye disorders) | 0 | 1 | 0
Periorbital edema (Eye disorders) | 0 | 0 | 0
Ptosis (Eye disorders) | 0 | 2 | 0
Retinopathy (Eye disorders) | 0 | 0 | 1
Vitreous hemorrhage (Eye disorders) | 0 | 0 | 1
Watering eyes (Eye disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 14 | 7 | 13
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 4 | 1 | 6
Bloody stool (Gastrointestinal disorders) | 1 | 0 | 2
Changes in teeth (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 70 | 18 | 36
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 76 | 45 | 74
Dry mouth (Gastrointestinal disorders) | 13 | 4 | 6
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 5
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 3
Esophagitis (Gastrointestinal disorders) | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 5 | 0 | 3
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 13 | 5 | 8
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 1 | 0
Hematochezia (Gastrointestinal disorders) | 0 | 0 | 2
Hemorrhoids (Gastrointestinal disorders) | 3 | 4 | 1
Irritable bowel syndrome NOS (Gastrointestinal disorders) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 4 | 0 | 1
Nausea (Gastrointestinal disorders) | 67 | 50 | 29
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 4 | 0 | 3
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 1 | 2
Sugar cravings (Gastrointestinal disorders) | 1 | 0 | 0
Tongue sensitivity (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 0 | 2
Typhlitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 33 | 22 | 16
Chills (General disorders) | 6 | 7 | 7
Diaphoresis (General disorders) | 3 | 2 | 7
Edema face (General disorders) | 6 | 3 | 2
Edema limbs (General disorders) | 40 | 14 | 20
Edema trunk (General disorders) | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 108 | 50 | 62
Fever (General disorders) | 17 | 9 | 21
Flu like symptoms (General disorders) | 7 | 12 | 10
Gait disturbance (General disorders) | 2 | 0 | 2
Infusion related reaction (General disorders) | 0 | 0 | 1
Injection site reaction (General disorders) | 1 | 0 | 0
Irritability (General disorders) | 2 | 0 | 1
Localized edema (General disorders) | 2 | 8 | 5
Malaise (General disorders) | 0 | 0 | 3
Non-cardiac chest pain (General disorders) | 4 | 2 | 7
Pain (General disorders) | 32 | 34 | 45
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder fistula (Hepatobiliary disorders) | 1 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 0 | 1
Liver abscess (Hepatobiliary disorders) | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 2 | 1
Autoimmune disorder (Immune system disorders) | 0 | 1 | 0
Lymphadenopathy (Immune system disorders) | 0 | 0 | 1
Seasonal allergies (Immune system disorders) | 0 | 0 | 2
Tongue swelling (Immune system disorders) | 0 | 0 | 1
Bladder infection (Infections and infestations) | 0 | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 4 | 5
C. difficile infection (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Ehrlichiosis (Infections and infestations) | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0
Foot infection (Infections and infestations) | 1 | 0 | 1
Gum infection (Infections and infestations) | 0 | 0 | 2
Infected cyst (Infections and infestations) | 1 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 5 | 3 | 8
Mucosal infection (Infections and infestations) | 3 | 0 | 1
Nail infection (Infections and infestations) | 1 | 2 | 3
Otitis media (Infections and infestations) | 1 | 2 | 2
Papulopustular rash (Infections and infestations) | 0 | 1 | 1
Parasitic infection NOS (Infections and infestations) | 0 | 0 | 1
Paronychia (Infections and infestations) | 2 | 0 | 0
Peripheral nerve infection (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pleural infection (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 2 | 1 | 0
Sinusitis (Infections and infestations) | 4 | 6 | 5
Skin infection (Infections and infestations) | 5 | 3 | 6
Small intestine infection (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Testicular infection (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 1 | 3
Upper respiratory infection (Infections and infestations) | 72 | 32 | 54
Urinary tract infection (Infections and infestations) | 7 | 4 | 6
Vaginal infection (Infections and infestations) | 1 | 0 | 2
Viral infection NOS (Infections and infestations) | 1 | 0 | 2
Wound infection (Infections and infestations) | 0 | 0 | 1
Yeast infection NOS (Infections and infestations) | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 7 | 8 | 8
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Chemical peel burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dog bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 8 | 7
Fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0
Patellar dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin wound NOS (Injury, poisoning and procedural complications) | 0 | 0 | 3
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tick bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tongue laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 39 | 14 | 31
Alkaline phosphatase increased (Investigations) | 18 | 7 | 14
Aspartate aminotransferase increased (Investigations) | 29 | 14 | 26
Blood bilirubin increased (Investigations) | 7 | 4 | 5
Cholesterol high (Investigations) | 0 | 2 | 1
Creatinine increased (Investigations) | 35 | 20 | 23
Elevated prostate antigen (Investigations) | 0 | 0 | 1
Fibrinogen decreased (Investigations) | 0 | 0 | 1
GGT increased (Investigations) | 2 | 0 | 0
Hemoglobin increased (Investigations) | 0 | 0 | 1
INR increased (Investigations) | 0 | 1 | 1
Lipase increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 144 | 47 | 60
Lymphocyte count increased (Investigations) | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 64 | 18 | 89
Platelet count decreased (Investigations) | 97 | 37 | 54
Serum amylase increased (Investigations) | 1 | 0 | 0
Transminitis NOS (Investigations) | 1 | 0 | 0
Weight gain (Investigations) | 8 | 3 | 2
Weight loss (Investigations) | 1 | 4 | 4
White blood cell decreased (Investigations) | 104 | 29 | 71
Anorexia (Metabolism and nutrition disorders) | 5 | 4 | 11
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 6 | 8 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 80 | 24 | 35
Hyperkalemia (Metabolism and nutrition disorders) | 8 | 8 | 9
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 15 | 6 | 9
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 4 | 4 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 23 | 1 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 30 | 5 | 20
Hypoglycemia (Metabolism and nutrition disorders) | 15 | 8 | 15
Hypokalemia (Metabolism and nutrition disorders) | 30 | 9 | 30
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 14 | 3 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 2 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 3
Achilles tendinosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 13 | 27
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 11 | 9
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 58 | 37 | 59
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 12 | 13
Bone spur (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 7 | 1 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 8 | 3 | 8
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 5 | 3
Gout (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hernia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Meniscus tear (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle cramps (Musculoskeletal and connective tissue disorders) | 13 | 7 | 23
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 14 | 28
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 14
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 31 | 30
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Tibialis anterior and EHL tendon laceration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Boil (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 5
Cystocele (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lump NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2
Mass NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nevi (benign) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 2
Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 2 | 1
Balance issues (Nervous system disorders) | 0 | 1 | 0
Concentration impairment (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 19 | 9 | 15
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 17 | 2 | 6
Dystonic reaction (Nervous system disorders) | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 1
Foot drop (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 23 | 8 | 21
Hypersomnia (Nervous system disorders) | 0 | 1 | 0
Left-sided numbness (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 3 | 1
Movements involuntary (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 9 | 6 | 12
Parkinsonism (Nervous system disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 12 | 9 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 89 | 48 | 65
Phantom pain (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Spinal stenosis (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 3 | 2 | 0
Tardive dyskinesia (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 6 | 1 | 4
Twitching (Nervous system disorders) | 2 | 0 | 0
Agitation (Psychiatric disorders) | 10 | 0 | 1
Anxiety (Psychiatric disorders) | 11 | 4 | 10
Confusion (Psychiatric disorders) | 3 | 4 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 1
Dementia (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 11 | 7 | 9
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 59 | 10 | 17
Psychosocial difficulties (Psychiatric disorders) | 0 | 1 | 0
Recurrent dreams (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 1
Bladder stones (Renal and urinary disorders) | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 4
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 1 | 3
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Renal calculi (Renal and urinary disorders) | 5 | 1 | 1
Urinary frequency (Renal and urinary disorders) | 5 | 3 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 2 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 4 | 4
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 1
Urostomy obstruction (Renal and urinary disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1 | 1
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 1 | 0 | 0
Premenstrual syndrome (Reproductive system and breast disorders) | 0 | 0 | 1
Prostate pain (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 4
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 27 | 46
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 32 | 20 | 27
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17 | 9 | 24
Nasal nares inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 8
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 11 | 5 | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Allergic contact dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Brittle nails (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Chalazion (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Chapped lips (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 5 | 17
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 4
Hypersensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ingrown toenail (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Laceration (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Poison ivy (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 6 | 7
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash NOS (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 33 | 24 | 27
Rosacea (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Roseola (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrheic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Shingles (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Skin hypersensitiviy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion NOS (Skin and subcutaneous tissue disorders) | 0 | 4 | 3
Skin tear NOS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Wart (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cataract surgery (Surgical and medical procedures) | 0 | 1 | 0
Crown dislodging (Surgical and medical procedures) | 1 | 0 | 0
Cyst removal (Surgical and medical procedures) | 0 | 0 | 1
Excision of lipoma (Surgical and medical procedures) | 0 | 0 | 1
Hernia repair (Surgical and medical procedures) | 0 | 0 | 1
Knee arthroscopy (Surgical and medical procedures) | 0 | 0 | 1
Knee replacement (Surgical and medical procedures) | 0 | 1 | 0
Oral surgery (Surgical and medical procedures) | 0 | 1 | 0
Orthopedic repair/surgery (Surgical and medical procedures) | 0 | 0 | 1
Root canal (Surgical and medical procedures) | 0 | 1 | 1
Spine surgery (Surgical and medical procedures) | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0
Flushing (Vascular disorders) | 6 | 1 | 0
Hematoma (Vascular disorders) | 0 | 0 | 2
Hot flashes (Vascular disorders) | 7 | 6 | 13
Hypertension (Vascular disorders) | 34 | 18 | 26
Hyperviscosity (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 10 | 4 | 4
Lymphedema (Vascular disorders) | 1 | 0 | 1
Superficial thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 5 | 1 | 6
Vascular calcification (Vascular disorders) | 0 | 0 | 1
Venous stasis (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT02253316/Prot_SAP_000.pdf